CLINICAL TRIAL: NCT02483143
Title: N-acetylcysteine, Sodium Bicarbonate and Normal Saline Alone Prophylaxis for Spiral Computed Tomography Pulmonary Angiography in the Emergency Department on Suspicion of Pulmonary Emboli: A Randomized Controlled Trial
Brief Title: NAC, NaHCO3 and NS Prophylaxis for CTPA in the ED on Suspicion of PE: A Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Suleyman Turedi, M.D., Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2014/47
Record Dates: First submitted 2015-05-27; First posted 2015-06-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Radiographic Contrast Agent Nephropathy; Pulmonary Embolism
Keywords: contrast media; pulmonary embolism; N-acetylcysteine
MeSH Terms: conditions — Pulmonary Embolism | interventions — Acetylcysteine; Sodium Bicarbonate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NAC plus normal saline group (Active Comparator): 1ml/3mgr NAC+NS preCTPA 3 ml/kg for 1 h, 1 ml/kg/h for post CTPA for 6 h
  Interventions: Drug: NAC
- NaHCO3 plus normal saline group (Active Comparator): 132 mEq NaHCO3+NS preCTPA 3 ml/kg for 1h, post CTPA 1ml/kg/h for 6 h
  Interventions: Drug: NaHCO3
- Normal saline alone (Placebo Comparator): preCTPA 3 ml/kg NS for 1h, postCTPA 1ml/kg/h SF for 6 h
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: NAC — 3 gr NAC was made up to 1000 ml with NS; a 1 ml/3 mgr NAC solution was obtained and 3 ml/kg NAC+NS solution was administered for 1 h before CTPA and a 1 ml/kg per hour NAC+NS solution was administered for a minimum 6 h after CTPA.
  Other Names: N-acetylcysteine
  Arms: NAC plus normal saline group
Drug: NaHCO3 — 132 mEq NaHCO3 was made up to 1000 ml with NS; and 3 ml/kg NaHCO3+NS solution was administered for 1 h before CTPA and 1 ml/kg per hour NaHCO3+NS solution was administered for a minimum of 6 h after CTPA.
  Other Names: Sodium Bicarbonate
  Arms: NaHCO3 plus normal saline group
Drug: Normal Saline — 3 ml/kg NS was administered for 1 h before CTPA and 1 ml/kg per hour was administered for a minimum of 6 h after CTPA.
  Other Names: Serum physiologic
  Arms: Normal saline alone

SUMMARY:
Study objective:

The purpose of this study was to compare the role of the prophylactic protocols N-acetylcysteine (NAC) plus normal saline, sodium bicarbonate (NaHCO3) plus normal saline and intravenous normal saline (NS) alone in the prevention of contrast-induced nephropathy (CIN) after computed tomography pulmonary angiography (CTPA) in emergency patients with suspected pulmonary embolism (PE).

Materials and methods:

This study was planned as randomized, double blind, placebo controlled clinical research. Patients presenting to the emergency department within a 1-year period, undergoing CTPA on suspicion of PE and having one or more risk factors for development of CIN were included in the study. The NAC group received 1 ml/3 mgr NAC+NS solution 1 h before CTPA and 1 ml/kg per hour for a minimum 6 h after CTPA. The NaHCO3 group received 132 mEq NaHCO3+NS solution for 1 h before CTPA and 1 ml/kg per hour for a minimum of 6h after CTPA. The normal saline (NS) group received 3 ml/kg NS for 1 h before CTPA and 1 ml/kg per hour NS for a minimum 6 h after CTPA. CIN was evaluated as the primary outcome, and moderate renal injury (defined as a 100% increase in serum creatinine levels), severe renal insufficiency requiring hemodialysis or peritoneal dialysis) or in-hospital mortality as secondary outcomes.

DETAILED DESCRIPTION:
Study Design and Setting This randomized, double blind, placebo control study was performed in the emergency department of a tertiary care university hospital in Turkey receiving >100,000 patient presentations annually. Approval was granted by the Karadeniz Technical University institutional ethical committee. Written and informed consent was received from all patients enrolled. The data collected period commenced on 1 February 2014, and the study period lasted for 1 year until 1 February 2015.

Selection of Participants Patients undergoing contrast enhanced thoracic tomography due to suspected PE, aged over 18, with measureable basal creatinine levels pre-tomography and measurable serum creatinine levels 48-72 h post-tomography and with one or more of the risk factors for CIN cited below were enrolled. The risk factors were pre-existing renal dysfunction (Cre 1.4 mg/dl or a high or calculated glomerular filtration rate <60 ml/min/1.73 m2), diabetes mellitus, hypertension receiving treatment, hypotension (SBP<90 mmHg), coronary artery disease, history of nephrotoxic drug use (NSAID, cisplatin, aminoglycoside, amphotericin B), liver disease, congestive heart failure (active or history thereof), age 65 or over, and anemia (Htc <30%). Patients refusing to participate or to provide informed consent, end stage renal patients already in peritoneal dialysis or hemodialysis, pregnant women, subjects with a known allergy to N-acetylcysteine or Na-bicarbonate, patients requiring NAC therapy or Na-bicarbonate therapy for existing additional disease, and patients exposed to contrast material for any reason in the previous 2 days were excluded. In addition, if the study protocol was considered by the physician responsible for treatment in the emergency department as being liable to delay medical care or have adverse effects, or if any of the drugs in the protocol were thought to be contraindicated, such patients were also excluded.

Interventions Computer-based block randomization was employed to randomize subjects. Three groups, A, B and C were established, each representing a drug branch treatment code.

The diagnostic approach algorithm to be applied in patients with suspected PE and the planning of treatment of PE were based on the 2014 ESC Guidelines on the diagnosis and management of acute pulmonary embolism.

In the NAC group; 3 gr NAC was made up to 1000 ml with NS; a 1 ml/3 mgr NAC solution was obtained and 3 ml/kg NAC+NS solution was administered for 1 h before CTPA and a 1 ml/kg per hour NAC+NS solution was administered for a minimum 6 h after CTPA. In the NaHCO3 group; 132 mEq NaHCO3 was made up to 1000 ml with NS; and 3 ml/kg NaHCO3+NS solution was administered for 1 h before CTPA and 1 ml/kg per hour NaHCO3+NS solution was administered for a minimum of 6 h after CTPA. In the NS group: 3 ml/kg NS was administered for 1 h before CTPA and 1 ml/kg per hour was administered for a minimum of 6 h after CTPA.

Clinical follow-up Post-CTPA prophylactic infusion was maintained for at least 6 h. Patients unable to complete that period were removed from the study and not included in the analysis.

Patients were regularly observed by the physician responsible for patient monitoring and by authors blind to the prophylactic alternatives received throughout the study. Creatinine measurements required for determining CIN development in 48 to 72 h were performed in the departments in which patients were hospitalized, while discharged patients were invited to return to the emergency department where venous blood specimens were collected using phlebotomy.

Outcome Measures CIN development (an increase ≥25% or 0.5 mg/dl in creatinine levels 48-72 h after contrast exposure compared to basal levels) was evaluated as the primary outcome in the study.

A secondary outcome was assessed as moderate renal injury developing during hospitalization (defined as a 100% increase in serum creatinine levels, severe renal failure requiring hemodialysis or peritoneal dialysis) or in-hospital mortality. Patients were monitored throughout hospitalization until either discharge or mortality.

ELIGIBILITY:
Inclusion criteria:

1. Patients undergoing contrast enhanced thoracic tomography due to suspected PE
2. aged over 18 years old
3. Measureable basal creatinine levels pre-tomography and measurable serum creatinine levels 48-72 h post-tomography
4. with one or more of the risk factors for CIN cited below were enrolled.

The risk factors were pre-existing renal dysfunction (Cre 1.4 mg/dl or a high or calculated glomerular filtration rate <60 ml/min/1.73 m2), diabetes mellitus, hypertension receiving treatment, hypotension (SBP<90 mmHg), coronary artery disease, history of nephrotoxic drug use (NSAID, cisplatin, aminoglycoside, amphotericin B), liver disease, congestive heart failure (active or history thereof), age 65 or over, and anemia (Htc <30%).

Exclusion criteria:

1. Patients refusing to participate or to provide informed consent
2. End stage renal patients already in peritoneal dialysis or hemodialysis
3. Pregnant women
4. Subjects with a known allergy to N-acetylcysteine or Na-bicarbonate
5. Patients requiring NAC therapy or Na-bicarbonate therapy for existing additional disease
6. Patients exposed to contrast material for any reason in the previous 2 days were excluded.
7. If the study protocol was considered by the physician responsible for treatment in the emergency department as being liable to delay medical care or have adverse effects, or if any of the drugs in the protocol were thought to be contraindicated, such patients were also excluded.
8. Patients unable to receive post-CT infusion for a minimum of 6 h were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Contrast induced nephropathy (CIN) development | Post contrast 48-72 hour
  An increase ≥25% or 0.5 mg/dl in creatinine levels 48-72 h after contrast exposure compared to basal levels

SECONDARY OUTCOMES:
moderate renal injury developing | up to 4 weeks, participants were followed for the duration of hospital stay, an expected average of 4 weeks
  Number of participants who have 100% increase in serum creatinine levels
severe renal failure developing | up to 4 weeks, participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Number of participants who require hemodialysis or peritoneal dialysis for the duration of hospital stay
in-hospital mortality | up to 4 weeks, participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Number of participants who die in the duration of hospital stay hospital. Patients were monitored throughout hospitalization until either discharge or mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Suleyman Turedi, Assoc.Prof., Principal Investigator — Karadeniz Technical University Faculty of Medicine
Locations (1):
- Karadeniz Technical University Faculty of Medicine, Trabzon, Turkey (Türkiye)

REFERENCES:
- [Derived] Turedi S, Erdem E, Karaca Y, Tatli O, Sahin A, Turkmen S, Gunduz A. The High Risk of Contrast-induced Nephropathy in Patients with Suspected Pulmonary Embolism Despite Three Different Prophylaxis: A Randomized Controlled Trial. Acad Emerg Med. 2016 Oct;23(10):1136-1145. doi: 10.1111/acem.13051. Epub 2016 Sep 27. PMID 27411777